CLINICAL TRIAL: NCT00780819
Title: Does Borderzone Contrast Enhancement on Intraoperative MRI During High Grade Glioma Resection Correlate With Residual Tumor?
Brief Title: Borderzone Sampling
Acronym: BZS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MEC 07-2-039; ABR-17679
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: High Grade Glioma; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PoleStar N20 intraoperative MRI (Experimental): PoleStar N20 intraoperative MRI
  Interventions: Device: PoleStar N20 intraoperative MRI

INTERVENTIONS:
Device: PoleStar N20 intraoperative MRI — low field strength mobile intraoperative MRI system (0,15 Tesla) with local Faraday shielding (using the StarShield system)
  Other Names: manufactured by Odin Medical Technologies (Yokneam, Israel), incorporated in Medtronic Navigation (Louisville, CO; USA)

SUMMARY:
On regular (diagnostic) MRI images brain tumors can show "contrast enhancement": uptake of an intravenously administered contrast agent can cause an enhancement pattern that is seen as a white area on a frequently used MRI protocol ("T1 weighted imaging"). High grade gliomas are a common brain tumor that share this enhancement pattern. The goal of surgery is to resect this contrast enhancing part without causing additional neurological damage. Intraoperative MRI (iMRI) is a helpful tool in achieving this goal, because it can provide updated images during resection and correct for deformations that occur in the brain during surgery. These deformations make preoperative images that are used for standard neuronavigation systems less reliable. However, due to manipulations during surgery, the contrast uptake during surgery may differ from contrast uptake in diagnostic MRI. This study aims to relate contrast enhancement on iMRI and tumor characteristics on tissue samples from the tumor. When the neurosurgeon considers the resection of the high grade glioma to be complete, an iMRI scan will be made, and tissue sampling will be performed on the borderzones of the tumor or tumor resection cavity respectively. This will provide insight in the relation between contrast enhancement on iMRI and the presence of tumor tissue. Such knowledge is important to improve effectiveness and safety of iMRI guided brain tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* supratentorial brain tumor, on contrast enhanced MRI suspect for a high grade glioma
* indication for resection of the tumor
* age ≥ 18 years
* WHO Performance Scale ≤ 2
* ASA class ≤ 3
* good knowledge of the Dutch language
* informed consent

Exclusion Criteria:

* recurrent tumor
* multiple tumor localizations
* prior radiotherapy on the skull
* prior chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The relation between the shape and size of contrast enhancement on intraoperative MRI at the resection cavity border, and the presence of residual tumor tissue. | after surgery, and after 1 year for additional immunochemistry

SECONDARY OUTCOMES:
The relation between possible contrast enhancement and contrast enhancing tissue volume on the last intraoperative MRI scan and the early diagnostic MRI scan | within 72 hours after surgery
Postoperative clinical condition (WHO Performance Scale) | 1 week after surgery
Survival (Kaplan Meier) | after 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Pieter L Kubben, MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands